CLINICAL TRIAL: NCT05342792
Title: Metronomic Capecitabine With or Without Tislelizuamb (PD-1 Antibody) as Adjuvant Therapy in High-risk Non-metastatic Nasopharyngeal Carcinoma: a Multicentre, Open-label, Randomised Phase 3 Trial
Brief Title: Metronomic Capecitabine With or Without PD-1 Antibody as Adjuvant Therapy in High-risk Nasopharyngeal Carcinoma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Tongji Hospital (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Xiangya Hospital of Central South University (Other); Affiliated Cancer Hospital of Guizhou Medical University (Unknown); Cancer Hospital of Guangxi Medical University (Other); First People's Hospital of Foshan (Other); Chongqing University Cancer Hospital (Other); Hubei Cancer Hospital (Other); Hunan Cancer Hospital (Other); The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); Fifth Affiliated Hospital, Sun Yat-Sen University (Other); Shandong Provincial Hospital (Other Government)
Responsible Party: Principal Investigator, Jun Ma, MD, Hospital Deputy Dean, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SL-B2022-202-02
Record Dates: First submitted 2022-04-17; First posted 2022-04-25 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: PD-1 antibody; Metronomic capecitabine; Adjuvant therapy
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — spartalizumab; tislelizumab; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metronomic Capecitabine with PD-1 antibody arm (Experimental): Patients randomised to this arm will receive metronomic capecitabine (650mg/m2, BID, PO) and Tislelizuamb (200mg, iv drip, Q3W) for 1 year as adjuvant therapy, beginning 4-6 weeks after chemoradiation.
  Interventions: Drug: PD-1 antibody; Drug: Capecitabine
- Metronomic Capecitabine alone arm (Active Comparator): Patients randomised to this arm will receive metronomic capecitabine (650mg/m2, BID, PO) alone for 1 year as adjuvant therapy, beginning 4-6 weeks after chemoradiation.
  Interventions: Drug: Capecitabine

INTERVENTIONS:
Drug: PD-1 antibody — Tislelizumab：200 mg per dose, intravenous infusion over 30 minutes, every 3 weeks as a cycle for 17 cycles after concurrent chemoradiotherapy
  Other Names: Tislelizumab
  Arms: Metronomic Capecitabine with PD-1 antibody arm
Drug: Capecitabine — Capecitabine : 650 mg/m2 bid, orally, d1-21, every 3 weeks as a cycle for 17 cycles after concurrent chemoradiotherapy

SUMMARY:
This trial is aimed to investigate whether additional adjuvant PD-1 antibody treatment could improve survival in high-risk nasopharyngeal carcinoma compared to metronomic capecitabine alone.

DETAILED DESCRIPTION:
In this multicenter, randomised controlled, phase 3 trial, patients with T4N+/TanyN2-3 (AJCC/UICC 8th system), or non-metastatic nasopharyngeal carcinoma with pretreatment EBV DNA > 4000 copies/ml, will be randomized in a 1:1 ratio to receive metronomic capecitabine with or without PD-1 antibody every 3 weeks for 1 year after curative chemoradiation.

ELIGIBILITY:
Inclusion Criteria:

1. Age at diagnosis: 18 ~ 65 years old;
2. Pathologically confirmed primary nasopharyngeal carcinoma with "non-keratinizing carcinoma (WHO criteria)";
3. Locoregionally advanced nasopharyngeal carcinoma (T4N + or TanyN2-3M0, or TanyNanyM0 pretreatment EBVDNA ≥ 4000 copies/mL) was diagnosed according to the American Joint Committee on Cancer/Union for International Cancer Control (AJCC/UICC) 8th edition clinical staging system.
4. Induction and concurrent chemoradiotherapy with the recommended regimen have been completed;
5. ECOG score: 0 ~ 1 points (Appendix II);
6. It is recommended to initiate adjuvant therapy within 1 month after the completion of the last radiotherapy treatment, no later than 6 weeks;
7. Normal bone marrow function: white blood cell count > 4 × 109/L, hemoglobin concentration > 90 g/L, platelet count > 100 × 109/L;
8. Normal liver and kidney function: total bilirubin ≤ 1.5 times the upper limit of normal; aspartate aminotransferase and/or alanine aminotransferase ≤ 2.5 times the upper limit of normal; alkaline phosphatase ≤ 2.5 times the upper limit of normal; creatinine clearance ≥ 60 mL/min;
9. Subjects must sign the informed consent form, and must be willing and able to comply with the visits, treatment regimen, laboratory tests and other requirements specified in the study protocol;
10. Female subjects of childbearing potential and male subjects with partners of childbearing potential must agree to use reliable contraception (e.g., condoms, regular contraceptives as directed) from screening through 1 year after treatment.

Exclusion Criteria:

1. Positive hepatitis B surface antigen and hepatitis B virus quantification > 1 × 1000 copies/ml, or positive anti-hepatitis C virus antibody;
2. Positive anti-HIV antibody or diagnosis of acquired immunodeficiency syndrome (i.e., AIDS);
3. Conditions such as dysphagia, chronic diarrhea, or bowel obstruction that would interfere with oral medication.
4. Patients with severe chronic or active infection that must be treated with systemic antibacterial, antifungal or antiviral therapy before randomization, including but not limited to tuberculosis infection
5. Active, known or suspected autoimmune disease (including but not limited to uveitis, enteritis, hepatitis, pituitary disease, nephritis, vasculitis, hyperthyroidism, hypothyroidism, and asthma requiring bronchiectasis). Except for type I diabetes, hypothyroidism requiring hormone replacement therapy and skin diseases not requiring systemic treatment (such as vitiligo, psoriasis or alopecia); clinicians should perform necessary history, examination and examination before enrollment for the above diseases and then exclude them;
6. Interstitial lung disease or pneumonia requiring oral or intravenous steroid therapy within 1 year;
7. Definite clinical evidence of persistent local disease or distant metastasis after chemoradiotherapy;
8. Systemic hormonal or other immunosuppressive therapy with an equivalent dose of > 10 mg prednisone/day within 28 days prior to informed consent. Subjects with systemic sex hormone doses ≤ 10 mg prednisone/day or inhaled/topical corticosteroids may be included.
9. Uncontrolled heart disease, such as: 1) heart failure, NYHA level ≥ 2; 2) unstable angina; 3) history of myocardial infarction in the past year; 4) supraventricular arrhythmia or ventricular arrhythmia requiring treatment or intervention;
10. Pregnant or lactating women (pregnancy test should be considered for sexually active women of childbearing age);
11. Previous or current other malignancy other than adequately treated non-melanoma skin cancer, carcinoma in situ of the cervix, and papillary thyroid carcinoma;
12. Receipt of live vaccines within 30 days prior to the first course of tislelizumab;
13. History of organ transplantation;
14. Other conditions that may jeopardize patient safety or compliance as assessed by the investigator, such as serious illness (including psychiatric disorders) requiring prompt treatment, severely abnormal test results, and other family or social risk factors.
15. Patients who received surgical treatment, biological therapy, or immunotherapy during or before radiotherapy;
16. Patients who are receiving or are likely to receive other chemotherapy, biological therapy, or immunotherapy History of severe hypersensitivity to other monoclonal antibodies;
17. Chemotherapy or surgery (except diagnostic) of the primary tumor or lymph nodes before standard treatment.
18. History of radiation therapy prior to standard therapy (except for non-melanoma skin cancer).
19. Patients who are known to be intolerable or sensitive to any therapeutic agents.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 556 (Estimated)
Dates: Start 2022-04-17 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
failure-free survival | 3 years
  calculated from the date of randomisation to the date of locoregional failure, distant failure, or death from any cause, whichever occurred first

SECONDARY OUTCOMES:
overall survival | 5 years
  calculated from date of randomisation to death
distant metastasis-free survival | 3 years
  calculated from date of randomisation to the first distant failure
locoregional recurrence-free survival | 3 years
  locoregional recurrence-free survival
adverse events (AEs) and severe adverse events (SAE) | 5 years
  graded according to NCI CTCAE v5.0
quality of life (QoL) | 3 years
  the change of QoL from randomization to 12 months after chemoradiation, graded according to EORTC QLQ-C30 V3.0

CONTACTS AND LOCATIONS:
Overall Officials: Jun Ma, MD, Principal Investigator — Sun Yet-senU
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
Complete de-identified patient data set
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 24 months following article publication
Access Criteria: Proposals should be emailed to the PI to gain access